CLINICAL TRIAL: NCT06806397
Title: Studying the Mechanisms of Visual-motor Transformation to Find Neurophysiological Markers of Altered Functions of Cortical Motor Circuits in Patients with Neurological Disorders and Developing Technologies for Their Rehabilitation.
Brief Title: Study of Hemodynamic Markers of Upper Extremity Motor Dysfunction in Stroke Patients Using Functional Near Infrared Spectroscopy (fNIRS)
Status: Recruiting | Type: Observational
Sponsor: Skolkovo Institute of Science and Technology (Other)
Collaborators: Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency of Russia (Unknown)
Responsible Party: Sponsor
Other Study IDs: Skoltech-CNBR7; 21-75-30024 (Other Grant/Funding Number: Russian Science Foundation)
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Stroke with Hemiparesis; Stroke, Ischemic
Keywords: stroke; hemiparesis; hemodynamics; fNIRS; restoration of motor function; Neurovascular coupling
MeSH Terms: conditions — Stroke; Ischemic Stroke; Paresis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals after stroke
  Interventions: Diagnostic Test: Stimulus response task
- Healthy volunteers
  Interventions: Diagnostic Test: Stimulus response task

INTERVENTIONS:
Diagnostic Test: Stimulus response task — Participants were tasked with performing a finger extension exercise that required pressing buttons in response to visual stimuli. In cases where physical movement was not possible, participants were instructed to imagine performing the task while focusing on their fingers.

SUMMARY:
The aim of the study was to explore potential pathways for recovery and adaptation of the motor cortex by examining cerebral blood flow characteristics and hemodynamic markers analyzed by functional near-infrared spectroscopy (fNIRS) in patients with hemiparesis after stroke. Participants in the study performed a simple stimulus-response task several times with one healthy and one paralyzed limb at different stages of basic rehabilitation. A group of healthy, age-matched volunteers participated in the same experiment to verify the stroke-related changes. The researchers recorded fNIRS signals, muscle activity using electromyography, and heart activity using electrocardiography.

DETAILED DESCRIPTION:
The study included 40 participants, divided into two groups: individuals with a history of stroke-related hemiparesis and a matched healthy control group.Participants were instructed to perform a stimulus-response task designed to assess reaction speed.During the task, they positioned their hands within a designated box equipped with two buttons corresponding to left and right responses. A visual stimulus, presented via LEDs located above the buttons, served as the response target. A flash of a stimulus required participants to respond by extending their fingers to press the corresponding button. If limb paresis prevented a full button press, participants were instructed to form an intention to move and attempt the task to the best of their ability.

Neurophysiological data acquisition. Functional near-infrared spectroscopy (fNIRS) data were acquired using a combined NIRSport 16x16 and NIRSport 8x8 system (NIRx Medizintechnik GmbH, Berlin, Germany).Twenty-four sources and 24 detectors were placed over the sensorimotor area and adjacent regions, forming 76 source-detector pairs to ensure comprehensive cortical coverage. The light sources were activated synchronously, resulting in a sampling rate of 13.56 Hz. In addition, surface electromyography (EMG), electrocardiography (ECG), and scalp electroencephalography (EEG) were recorded using the NVX-36 electroencephalograph (ISS, Zelenograd, Russia). EMG activity was recorded from the extensor digitorum communis muscle of both hands using a bipolar belly-tendon montage. ECG was recorded by 1st standard bipolar montage with electrode placed on both wrists. EEG was recorded with 6 electrodes placed at 'FCC3', 'FCC4', 'CCP3', 'CCP4', 'FCC5', 'A1', 'FCC6', 'A2' according to the standard "10-05" montage. The experimental protocol was completed within two weeks for each participant. There were six sessions (3 at the beginning of rehabilitation and 3 before discharge). Each session lasted a maximum of one hour. Before the experimental session, each patient's motor abilities were tested using the Action Research Arm Test (ARAT) and the Fugl-Meyer Assessment (FMA) scale.

ELIGIBILITY:
For Healthy Volunteers:

Inclusion Criteria:

1. Availability of signed written informed consent. 3. Absence of somatic and psychiatric diseases (more details in the exclusion criteria) 4. Ability and willingness to comply with the requirements of this protocol.

Exclusion Criteria:

1. The presence of superficial injury of head (S00-S09 International Classification of Diseases 10 (ICD-10).
2. The presence of mental, behavioural disorders (F00-F99 ICD-10).
3. Drug addiction in the past or at the moment.
4. The presence of diseases of the nervous system (G00-G99 ICD-10).
5. . History of intracranial injury (S06 ICD-10) or stroke (I64 ICD-10).
6. The presence of somatoform disorders (F45 ICD-10).
7. Any conditions that, in the opinion of the Investigator, meet the exclusion criteria
8. Presence of electrical and/or metallic implants or stimulants in the body (eg, implanted deep brain stimulation devices, pacemakers, hearing aids and cochlear implants, intracranial metal implants).
9. Pregnancy
10. The presence of malignant neoplasms (C00-C97 ICD-10).

For stroke patients:

Inclusion Criteria:

1. Signed written informed consent.
2. People after the first acute cerebrovascular accident (CVA), early or late rehabilitation period.
3. The level of severity of paresis of the upper limb from 3 points to 0 (according to a 6-point neurological scale)
4. The minimum visual acuity is not lower than 0.2 on the Sivtsev scale.
5. The ability and willingness of the patient to comply with the requirements of this protocol.
6. Expressed patient motivation for rehabilitation.

Exclusion Criteria:

1. Severe cognitive impairment (<10 points according to the Montreal Cognitive Assessment Scale).
2. Hamilton score above 18 points.
3. The score on the Rankin scale is above 4 points.
4. Associated neurological disorders that cause decreased muscle strength or increased muscle tone in the upper limbs (eg, cerebral palsy, brain damage from trauma) or stiffness (eg, Parkinson's disease, contracture).
5. Late stages of arthritis or clinically significant limitation of passive range of motion in any of the joints studied in the study due to other reasons.
6. The absence of a part of the upper limb due to amputation caused by various reasons.
7. Any medical condition, including mental illness or epilepsy, that may affect the interpretation of study results, study conduct, or patient safety.
8. Alcohol abuse, medical marijuana use, or recreational drug use in the 12 months prior to Visit 1.
9. Use of experimental drugs or medical devices within 30 days prior to Visit 1.
10. Lack of ability to follow study procedures, in the opinion of the investigator.
11. The severity of the patient's condition according to the neurological or somatic status, which does not allow full rehabilitation.
12. Severe visual disturbances, minimal visual acuity less than 0.2 Sivtsev visual acuity table.
13. Unstable angina and/or heart attack within the previous month
14. Repeated stroke.
15. Severe unilateral spatial neglect.
16. Uncontrolled arterial hypertension
17. Ataxia
18. All forms of epilepsy

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing rehabilitation at the Federal center of brain research and neurotechnologies, FMBA, Moscow, Russia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic changes after stroke | 14 days
  In post-stroke subjects, an increase in blood flow and oxygenation was observed in sensorimotor cortical regions of both hemispheres during movement of the paretic limb. This observation may indicate that the healthy hemisphere contributes to the execution of movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Skolkovo Institute of Science and Technology (Skoltech), Moscow, Russia